CLINICAL TRIAL: NCT04982913
Title: A Single-Center, Randomized, Double-Blind, Single and Multiple Doses, Placebo-Controlled Study,To Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics, Food Effects of HEC116094HCl•3H2O and the Interaction With Oseltamivir Phosphate Capsules in Chinese Healthy Subjects
Brief Title: Single Dose and Multiple Dose Safety, Tolerability, PK，and Food Effect Study，and Interaction With Oseltamivir Study of HEC116094 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HEC116094-P-01/CRC-C2104
Record Dates: First submitted 2021-07-23; First posted 2021-07-29 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Single dose of HEC116094（Part A, Cohort 1） (Experimental): Healthy subjects receive sinele dose of HEC116094
  Interventions: Drug: HEC116094
- Single dose of HEC116094（Part A, Cohort 2） (Experimental): Healthy subjects receive sinele dose of HEC116094 or matching placebo
  Interventions: Drug: HEC116094
- Single dose of HEC116094（Part A, Cohort 3） (Experimental): Healthy subjects receive sinele dose of HEC116094 or matching placebo
  Interventions: Drug: HEC116094
- Single dose of HEC116094（Part A, Cohort 4，Fed/Fasting） (Experimental): Following an overnight fast of at least 10 hours, a single dose of HEC116094 will be administered on 2 separate occasions (fasting and after meal) in a randomized crossover fashion with different food restrictions.
  Interventions: Drug: HEC116094
- Single dose of HEC116094（Part A, Cohort 5） (Experimental): Healthy subjects receive sinele dose of HEC116094 or matching placebo
  Interventions: Drug: HEC116094
- Single dose of HEC116094（Part A, Cohort 6） (Experimental): Healthy subjects receive sinele dose of HEC116094 or matching placebo
  Interventions: Drug: HEC116094
- Single dose of HEC116094（Part A, Cohort 7） (Experimental): Healthy subjects receive sinele dose of HEC116094 or matching placebo
  Interventions: Drug: HEC116094
- Mulltiple doses HEC116094（ Part B, Cohort 1） (Experimental): Healthy subjects receive multiple doses of HEC116094 or matching placebo
  Interventions: Drug: HEC116094
- Mulltiple doses HEC116094（ Part B, Cohort 2） (Experimental): Healthy subjects receive multiple doses of HEC116094 or matching placebo
  Interventions: Drug: HEC116094
- Mulltiple doses HEC116094（ Part B, Cohort 3） (Experimental): Healthy subjects receive multiple doses of HEC116094 or matching placebo
  Interventions: Drug: HEC116094
- Mulltiple doses HEC116094（ Part B, Cohort 4） (Experimental): Healthy subjects receive multiple doses of HEC116094 or matching placebo
  Interventions: Drug: HEC116094
- The interaction with Oseltamivir of HEC116094（ Part C） (Experimental): Healthy subjects received HEC116094 in cycle 1, Oseltamivir in cycle 2, and a combination of HEC116094 and Oseltamivir in cycle 3.There are washout periods between the first cycle and the second cycle and between the second cycle and the third cycle
  Interventions: Drug: HEC116094

INTERVENTIONS:
Drug: HEC116094 — Part B：Mulltiple doses up to 5 days； Part C：Each cycle was administered for 5 days
  Other Names: Oseltamivir

SUMMARY:
The Safety, Tolerability, Pharmacokinetic, Food Effect Study and the interaction with Oseltamivir Phosphate Capsules of HEC116094 in Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in the study, able to understand and sign the informed consent, and able to complete the the study in accordance with the requirements of the study.
* Female subjects who are not pregnant or lactating and male subjects whose female partners are fertile shall voluntarily take effective contraceptive measures from the date of signing the informed consent form to 3 months after the medication.
* When signing the informed consent, 18 years old ≤the age≤45 years old(including the critical value), gender is not limited.
* Male body weight ≥50kg, female body weight ≥45kg, and body mass index (BMI) in the range of 18-28 kg/m2 (including the critical value).
* No clinical significance of vital signs, physical examination, laboratory examination, electrocardiogram, ultrasound abdomen and chest X-ray (posterior and anterior) results.

Exclusion Criteria:

* Positive for Viral hepatitis (including hepatitis B and C), HIV and syphilis.
* Those who are known to have allergy history or allergy constitution to the test preparation and any of its components or related preparations.
* Consume foods or beverages containing caffeine, xanthine, alcohol, and grapefruit within 48 hours prior to initial dosing.
* Positive results from urine drug screen test.
* Donate blood or lose blood 400 mL or more within 1 month prior to initial dosing.
* Subjects who plan to receive or have had organ transplants.
* Subjects considered by the investigator to have other factors unsuitable for participation in this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2021-08-24 (Actual); Primary Completion 2022-10-02 (Actual); Study Completion 2022-10-02 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of HEC116094 by Assessment of the Number of Adverse | up to 7 days at Part A and 11 days at Part B and 26 days at Part C
  To investigate the safety and tolerability of HEC116094 by assessment of AEs

SECONDARY OUTCOMES:
Cmax | up to 72 hours
  Maximum Plasma Concentration(Cmax)of HEC116094
AUC | up to 72 hours
  Area Under the Curve(AUC) of HEC116094
Tmax | up to 72 hours
  Maximum Peak Time(Tmax) of HEC116094
T1/2 | up to 72 hours
  Maximum Peak Time(Tmax) of HEC116094

CONTACTS AND LOCATIONS:
Locations (1):
- The Shanghai xuhui district central hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No